CLINICAL TRIAL: NCT05659407
Title: The BAFF-var Polymorphism as a Biomarker of Response to B-depletive Treatment in Patients Affected by Systemic Lupus Erythematosus and Rheumatoid Arthritis: a Prospective Study
Brief Title: BAFF-var as a Biomarker of Response to B-depletive Treatment in Systemic Lupus Erythematosus and Rheumatoid Arthritis
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Ospedaliero Universitaria di Cagliari (Other)
Responsible Party: Principal Investigator, Matteo Piga, Prof., University of Cagliari
Other Study IDs: PREDICT-SLE/RA
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis; BLyS Polymorphism
Keywords: Systemic lupus Erythematosus; Rheumatoid Arthritis; BLyS Polymorphism; Belimumab; Rituximab
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — belimumab; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For BAFF genotyping, whole blood samples will be collected in EDTA at the enrollment. The gDNA will be extracted by the salting-out method according to standard protocol. Customs TaqMan assay specifically designed to genotype the BAFF variants of interest will be used with allele-specific Real Time PCR in all samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BAFF-var carrier
  Interventions: Drug: Belimumab in SLE patients / Rituximab in RA patients
- No BAFF-var carrier
  Interventions: Drug: Belimumab in SLE patients / Rituximab in RA patients

INTERVENTIONS:
Drug: Belimumab in SLE patients / Rituximab in RA patients — Belimumab and Rituximab are the the investigated treatments, respectively in the SLE and RA group. They are administrated according to the approved indications and in compliance with the current recommendations and the good clinical practice, independently to the aim of the present observational study.

SUMMARY:
A variant of the TNFSF13B gene, commonly referred to as BAFF-var has been associated with an increased risk of developing immune-mediated diseases, such as Systemic Lupus Erythematosus (SLE) and Rheumatoid Arthritis (RA).

This polymorphism leads to the production of higher levels of BAFFs, that in turns are associated with more severe disease, high anti-Sm and anti-dsDNA titre, complement consumption, and increased risk of flare in SLE, and higher disease activity in RA.

This is a prospective study aiming to explore the immunological basis of a potential role of BAFF-var as a prognostic biomarker for response to belimumab and rituximab, the main B-depletive treatments, in SLE and RA patients, respectively. More in detail, the study aims to evaluate if the condition of BAFF-var carrier in SLE and RA patients, treated respectively, with belimumab plus standard of care or rituximab influences immunological, molecular and clinical variables, such as: (a) soluble BAFF (BAFFs) cytokine, (b) mRNA-BAFF (c) miRNA-15a (d) B-cell subpopulations (d) disease activity, as assessed by standardized clinimetric tools.

DETAILED DESCRIPTION:
BACKGROUND

Systemic lupus erythematosus (SLE) and Rheumatoid Arthritis (RA) are multisystem immune-mediated disease characterized by a complex pathogenesis, where an abnormal activation of the humoral immune response, with overproduction of autoantibodies, demonstrated to have a pivotal role.

B lymphocyte stimulator (BAFF) is a cytokine and drug target that is primarily produced by monocytes and neutrophils. It is essential for B-cell activation, differentiation and survival. Overexpression of BAFF was demonstrated to be associated with more severe pattern of SLE and correlate to more frequent positivity for anti-Sm (OR 1.7; 95% CI 1.3, 2.2), high titre anti-dsDNA (OR 1.5; 95% CI 1.1, 2.2), lower C3 (OR 1.3; 95% CI 1.0, 1.8), higher proteinuria (OR 1.8; 95% CI 1.4, 2.4) and increased risk of flare (HR 1.86; 95% CI 1.29, 2.68). Similarly, high levels of BAFF have been observed in blood and synovial fluid of RA patients and were demonstrated to correlate with higher disease activity in RA.

Belimumab and rituximab are the prototypical form of B-cell targeted therapies currently approved for SLE and RA, respectively.

Belimumab, a fully humanized monoclonal antibody directed against BAFF, is the first biological drug licensed and approved for use in combination with standard immunosuppressants in SLE. Data from RCTs demonstrated that higher disease activity, anti-dsDNA positivity, low complement and corticosteroid treatment may predict a higher benefit to belimumab. However, around 40% of subjects did not achieve an adequate response.

Rituximab (RTX) is a chimeric monoclonal antibody that of selectively inhibit the CD20 receptor on the surface of B lymphocytes. The use of RTX, preferably in combination with methotrexate, is indicated in patients with RA unresponsive to treatment with traditional immunosuppressants. Although greater efficacy was recorded in patients with positivity for autoantibodies (e.g. rheumatoid factor and anti-citrullinated peptide), also in this case a about 30-40% of patients is inadequately responsive.

A variant of TNFSF13B gene encoding for BAFF (BAFF-var), especially common across Sardinia (allele frequency, 26.5%) and progressively less common in southern (5.7% in Italy, 5.0% in Spain and Portugal) and northern Europe (1.8% in the UK and Sweden), was associated with autoimmune diseases, including SLE and RA. The causal variant was identified as an insertion-deletion variant, yielding a shorter transcript that escaped microRNA inhibition and increased production of soluble BAFF, which in turn up-regulated humoral immunity. In particular, BAFF-var was associated with increased level of soluble BAFF (effect size 0.77 standard deviations (SD); P= 8.47 x10-150), IgG (0.31 SD, p=1.68x10-12), IgA (0.31 SD, p=7.64x10-9), IgM (0.31 SD, p=4.70x10-8), as well as increased number of total B cell (0.18 SD, P=4.23x10-12) and several subtypes, including the CD24+CD27+ (comprising un-switched and switched memory) (0.22 SD, P=2.94x10-10) as the strongly associated. Further, transcriptome data demonstrated BAFF-var as an expression quantitative trait locus that increases TNFSF13B expression (P = 2.37×10-13). However, the elevated mRNA levels could explain only 24-27% of the effect on protein, indicating that an increase in translation level was also probably involved. In this regard, data indicate that BAFF-var raises soluble BAFF levels by favoring the production of a shorter transcript that is less inhibited by microRNA, such as miR-15a6.

Knowing the effective influence of BAFF-var in the immunological, molecular and clinical modifications induced by BAFF-inhibition has a crucial importance In the prospective of a personalized medicine in SLE and RA patients.

OBJETVIES

* Primary objective: To explore the immunological basis of a potential role of BAFF-var as a prognostic biomarker for response to belimumab or rituximab in the treatment SLE and RA patients, respectively. More in detail, the study aims to evaluate if the condition of BAFF-var carrier influences the drug-related modifications of immunological and molecular variables, such as: (a) soluble BAFF (BAFFs) cytokine, (b) mRNA-BAFF (c) miRNA-15a (d) B-cell subpopulations.
* Secondary objectives: To explore the effect of BAFF-var on the clinical response rate to belimumab or rituximab, as assessed by different outcome measures.

RESEARCH DESIGN AND METHODOLOGY

* Study design: The proposed project is an observational longitudinal study
* Population: Distribution of BAFF-var and modifications on immunological, molecular and clinical variables, after starting treatment with anti-BAFF agent, will be analyzed on a real-life monocentric Sardinian cohort of SLE and RA patients. In this regard, the Sardinian represents the most suitable population for this kind of analysis because of the higher frequency of BAFF-var; indeed the condition of BAFF-var carrier is expected in 50-60% of patients. About 30 consecutive SLE and 30 consecutive RA patents referred to the Rheumatology Unit at the Department of Medical Sciences and Public Heath of the University and University Clinic of Cagliari will be recruited.
* Data collection: Demographic (e.g. gender, age at enrolment, age of onset and diagnosis), clinical (e.g. cumulative and active disease manifestations, clinimetric measures), serological (e.g. autoantibodies, including anti-dsDNA, C3 and C4, IgG, IgA, IgM, RF, ACPA) and therapeutic (e.g past and current therapies) will be collected.
* BAFF genotyping: For BAFF genotyping, whole blood samples will be collected in EDTA at the enrollment. The gDNA will be extracted by the salting-out method according to standard protocol. Customs TaqMan assay (Thermo Fisher Scientific) specifically designed to genotype the BAFF variants of interest will be used with allele-specific Real Time PCR in all samples.
* B-cell phenotyping: Flow cytometry will be used to profile B-cell subpopulations in the 30 enrolled SLE patients. The number of B cell (CD45+CD19+), as well as the absolute and relative number of B transitional (CD24+CD38+), antibody secreting (ASC, CD27+CD38+), B memory switched (CD27+IgD-), B memory un-switched (CD27+IgD+), B naïve (IgD+CD27-CD24-) and B regulatory (CD24+CD27+) cells will be assessed by Lyse-No-Wash protocol using BD TruCountTM (Becton Dickinson).
* Soluble BAFF: it will be measured by enzyme-linked immunosorbent assay (ELISA)
* Gene expression study: mRNA will be extracted from whole blood by Trizol Reagent and the quantitative analysis of mRNA-BAFF and miRNA-15a will be performed by Real-Time PCR using specific TaqMan probes, after reverse transcription in cDNA.
* Statistical analysis. Statistical analysis will be performed by using the SPSS® statistical software. Comparison of mean levels of sBAFF, mRNA-BAFF, miRNA-15a and different B-cell phenotypes between BAFF-var + and BAFF-var - patients at each visit will be performed by T- Student test or Mann Whitney test, if appropriate. Comparison of the mean difference of levels of sBAFF, mRNA-BAFF, miRNA-15a and B-cell subpopulations between BAFF-var + and BAFF-var - patients at the different visits intervals will be performed by T- Student test or Mann Whitney test, if appropriate. The effect of BAFF-var on modification of the levels of the immunological and molecular variables above will be further assessed by multiple regression, including as independent variables, concomitant treatments and baseline disease features. Fisher's exact test and logistic regression analysis will be performed to compare the response rate, as assessed by different efficacy measures, in BAFF-var + and BAFF-var - patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* SLE diagnosis according to the '97 ACR Criteria / RA diagnosis to the ACR/EULAR 2010 criteria
* Belimumab / Rituximab initiation at the enrollment, according to the product indications.
* Treatment with glucocorticoids stable over the previous 4 weeks
* Treatment with other immunosuppressant stable over the previous 12 weeks

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A real-life monocentric cohort of consecutive patients affected by SLE and RA (recruited in the Rheumatology Unit, University Clinic of Cagliari), who started treatment with, respectively, belimumab or rituximab at the enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
BAFFs | 12 months
  Comparison of BAFFs level before and after treatment in BAFF-var carrier and no BAFF-var carrier
mRNA-BAFF e miRNA-15a | 12 months
  Comparison of mRNA-BAFF e miRNA-15a levels before and after treatment in BAFF-var carrier and no BAFF-var carrier
B-cell subpopulations | 12 months
  B-cell phenotyping before and after treatment in BAFF-var carrier and no BAFF-var carrier

SECONDARY OUTCOMES:
Delta PGA in SLE patients | 12 months
  Comparison of Physician Global Assessment of disease activity (PGA) on a VAS scale before and after treatment in BAFF-var carrier and no BAFF-var carrier
SLE responder index (SRI) in SLE patients | 12 months
  defined by a 4-point reduction in SELENA-SLEDAI score, no new BILAG A organ domain score and ≤ 1 new BILAG B score, and no increase ≥ 0.3 in PGA score vs. baseline;
Achievement of clinical remission ins SLE patients | 12 months
  Defined by SLEDAI-2k=0, PGA ≤ 0.5, prednisone (or equivalent) dosage ≤ 7.5mg daily
Delta PGA in RA patients | 12 months
  Comparison of Physician Global Assessment of disease activity (PGA) on a VAS scale before and after treatment in BAFF-var carrier and no BAFF-var carrier
Delta DAS-28 in RA patients | 12 months
  Comparison of DAS 28 before and after treatment in BAFF-var carrier and no BAFF-var carrier
EULAR response in RA patients | 12 months
  Response to treatment according to the EULAR criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Piga, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent FB, Morand EF, Schneider P, Mackay F. The BAFF/APRIL system in SLE pathogenesis. Nat Rev Rheumatol. 2014 Jun;10(6):365-73. doi: 10.1038/nrrheum.2014.33. Epub 2014 Mar 11. PMID 24614588
- [Background] Wei F, Chang Y, Wei W. The role of BAFF in the progression of rheumatoid arthritis. Cytokine. 2015 Dec;76(2):537-544. doi: 10.1016/j.cyto.2015.07.014. Epub 2015 Jul 18. PMID 26198030
- [Background] Petri MA, van Vollenhoven RF, Buyon J, Levy RA, Navarra SV, Cervera R, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Baseline predictors of systemic lupus erythematosus flares: data from the combined placebo groups in the phase III belimumab trials. Arthritis Rheum. 2013 Aug;65(8):2143-53. doi: 10.1002/art.37995. PMID 23754628
- [Background] Petri M, Stohl W, Chatham W, McCune WJ, Chevrier M, Ryel J, Recta V, Zhong J, Freimuth W. Association of plasma B lymphocyte stimulator levels and disease activity in systemic lupus erythematosus. Arthritis Rheum. 2008 Aug;58(8):2453-9. doi: 10.1002/art.23678. PMID 18668552
- [Background] Manzi S, Sanchez-Guerrero J, Merrill JT, Furie R, Gladman D, Navarra SV, Ginzler EM, D'Cruz DP, Doria A, Cooper S, Zhong ZJ, Hough D, Freimuth W, Petri MA; BLISS-52 and BLISS-76 Study Groups. Effects of belimumab, a B lymphocyte stimulator-specific inhibitor, on disease activity across multiple organ domains in patients with systemic lupus erythematosus: combined results from two phase III trials. Ann Rheum Dis. 2012 Nov;71(11):1833-8. doi: 10.1136/annrheumdis-2011-200831. Epub 2012 May 1. PMID 22550315
- [Background] Cohen SB, Emery P, Greenwald MW, Dougados M, Furie RA, Genovese MC, Keystone EC, Loveless JE, Burmester GR, Cravets MW, Hessey EW, Shaw T, Totoritis MC; REFLEX Trial Group. Rituximab for rheumatoid arthritis refractory to anti-tumor necrosis factor therapy: Results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial evaluating primary efficacy and safety at twenty-four weeks. Arthritis Rheum. 2006 Sep;54(9):2793-806. doi: 10.1002/art.22025. PMID 16947627
- [Background] Steri M, Orru V, Idda ML, Pitzalis M, Pala M, Zara I, Sidore C, Faa V, Floris M, Deiana M, Asunis I, Porcu E, Mulas A, Piras MG, Lobina M, Lai S, Marongiu M, Serra V, Marongiu M, Sole G, Busonero F, Maschio A, Cusano R, Cuccuru G, Deidda F, Poddie F, Farina G, Dei M, Virdis F, Olla S, Satta MA, Pani M, Delitala A, Cocco E, Frau J, Coghe G, Lorefice L, Fenu G, Ferrigno P, Ban M, Barizzone N, Leone M, Guerini FR, Piga M, Firinu D, Kockum I, Lima Bomfim I, Olsson T, Alfredsson L, Suarez A, Carreira PE, Castillo-Palma MJ, Marcus JH, Congia M, Angius A, Melis M, Gonzalez A, Alarcon Riquelme ME, da Silva BM, Marchini M, Danieli MG, Del Giacco S, Mathieu A, Pani A, Montgomery SB, Rosati G, Hillert J, Sawcer S, D'Alfonso S, Todd JA, Novembre J, Abecasis GR, Whalen MB, Marrosu MG, Meloni A, Sanna S, Gorospe M, Schlessinger D, Fiorillo E, Zoledziewska M, Cucca F. Overexpression of the Cytokine BAFF and Autoimmunity Risk. N Engl J Med. 2017 Apr 27;376(17):1615-1626. doi: 10.1056/NEJMoa1610528. PMID 28445677